CLINICAL TRIAL: NCT03471806
Title: Dopamine Release to Food Reward in Bulimia Nervosa: an [18F]-Fallypride PET/MR Study.
Brief Title: Dopamine Release to Food Reward in Bulimia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Associate Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S60362-BN
Record Dates: First submitted 2018-03-05; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Bulimia Nervosa; Food Reward
Keywords: Bulimia Nervosa; Eating disorder; Dopamine; Food; Reward; Positron Emission Tomography; Magnetic Resonance; Metabolic hormones
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulimia Nervosa patients (Experimental): Bulimia Nervosa patient group: Assessment of dopamine release to food reward at baseline (before treatment) and to food reward after treatment.
  Interventions: Behavioral: Food reward at baseline; Behavioral: Food reward after treatment
- Healthy controls (Experimental): Healthy control group: Assessment of dopamine release to food reward at baseline, for comparison with Bulimia Nervosa patients.
  Interventions: Behavioral: Food reward at baseline

INTERVENTIONS:
Behavioral: Food reward at baseline — Exposure to a combination of anticipatory (viewing high-calorie food images) and consummatory food reward (drinking sips of chocolate milkshake), at baseline.
Behavioral: Food reward after treatment — Exposure to a combination of anticipatory (viewing high-calorie food images) and consummatory food reward (drinking sips of chocolate milkshake), at the end of inpatient treatment.
  Arms: Bulimia Nervosa patients

SUMMARY:
This study will assess the role of dopamine responses to food reward in Bulimia Nervosa patients, by performing simultaneous Positron Emission Tomography (PET) and Magnetic Resonance (MR) scanning. The dopamine response will be measured before and after treatment, and will be compared to healthy controls.

DETAILED DESCRIPTION:
Bulimia nervosa is a psychiatric eating disorder characterized by recurrent episodes of binge eating, followed by inappropriate compensatory behaviour. It is associated with a high disease burden and high rates of medical and psychiatric comorbidities. Only 50% of patients achieve long-term remission, indicating the need for a better understanding of the pathophysiology which can guide the development of new treatment options.

There are strong indications for an involvement of the brain's dopaminergic reward system in Bulimia Nervosa, such as the presence of elevated craving for rewarding food and poorer impulse control. However, there is no clear evidence on the exact involvement of the reward system nor direct evidence of abnormal dopamine responses to food reward. Therefore, the current study will assess dopamine release and related brain activity to food reward in Bulimia Nervosa patients, by performing simultaneous Positron Emission Tomography (PET) and Magnetic Resonance (MR) scanning. Specifically, the investigators will compare dopamine release in Bulimia Nervosa patients to healthy controls, and assess the effect of successful treatment on the food reward response. To this end, 20 Bulimia Nervosa patients will participate in one PET-MR scan before the start of inpatient treatment and in a second PET-MR scan at the end of inpatient treatment. Additionally, PET-MR scans will be obtained from a group of 20 healthy control participants.

All scan session will measure dopamine release to a combination of anticipatory (viewing high-calorie food images) and consummatory (drinking sips of chocolate milkshake) food reward and will be conducted in a fasted state. The scan sessions will consist of four blocks with a duration of 45 minutes each and 15 minute breaks in between. The first three blocks represent the 'control condition' and the fourth block the 'food reward condition'. During both sessions, blood samples will be collected at several time points to assess levels of metabolic hormones and their relation to food-induced dopamine release.

This study aims to improve our understanding of the disease process underlying Bulimia Nervosa and to enable the identification of new and specific treatment targets at multiple levels of the gut-brain axis, including the dopamine system in the brain but also metabolic hormones and the interactions between both. Additionally, the results may have the potential to guide the optimisation of behavioural treatment approaches with a stronger focus on aberrant reward system responses.

ELIGIBILITY:
Patients with Bulimia Nervosa:

Inclusion Criteria:

* Diagnosed with Bulimia Nervosa based on DSM-5 criteria;
* Admission for inpatient treatment;
* Female (on hormonal contraception);
* Dutch-speaking;
* Right-handed;
* Body Mass Index (BMI) of 18.5 - 25 kg/m².

Exclusion Criteria:

* Medical, neurological or other psychiatric disorders;
* Use of psychotropic medication in past 6 months;
* Use of cannabis or other drugs of abuse in past 12 months;
* Lactose-intolerance or food allergies;
* Vegetarian diet;
* Smoking;
* Consumption of more than 7 alcoholic units per week;
* Exposure to a significant amount of ionizing radiation in past 12 months;
* Claustrophobia;
* Contra-indications for Magnetic Resonance Imaging;
* Pregnancy.

Healthy control participants:

Inclusion Criteria:

* Healthy females (on hormonal contraception);
* Dutch-speaking;
* Right-handed;
* Stable body weight with BMI of 18.5 - 25 kg/m².

Additional Exclusion Criteria:

* Any psychiatric disorders;
* Emotional or restraint eating behaviour.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Dopamine release to food reward in Bulimia Nervosa patients compared to healthy controls | Continuously over 225 minutes after onset scanning; at baseline (before onset treatment of patients)
  Comparison of dopamine release to food reward between Bulimia Nervosa patients and healthy controls. Dopamine release is defined as changes in [18F]-Fallypride binding potential in the food reward condition, with a kinetic linearized simplified reference region model (LSSRM) model.
Change in dopamine release to food reward in Bulimia Nervosa patients before and after treatment | Continuously over 225 minutes after onset scanning; before and after inpatient treatment
  Comparison of dopamine release to food reward before and after inpatient treatment for Bulimia Nervosa. Dopamine release is defined as changes in [18F]-Fallypride binding potential in the food reward condition, with a kinetic linearized simplified reference region model (LSSRM) model.

SECONDARY OUTCOMES:
Composite measure of metabolic hormone levels | 5 minutes before onset scanning and 45, 105, 165, 180, 195, 210 and 225 minutes after onset scanning
  Correlation between dopamine response to food reward and (changes in) metabolic hormone levels (ghrelin, motilin, glucagon-like peptide 1, peptide tyrosine tyrosine, leptin, and insulin)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, Prof. dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided